CLINICAL TRIAL: NCT06021600
Title: A Phase 1, Open-Label, Sequential Cross-over, Bioavailability/Bioequivalence Study to Compare the Pharmacokinetics of Oral Cladribine With the Reference Listed Drug, Intravenous Cladribine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0134; NCI-2023-06805 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Pilot) (Experimental): Participants will only receive 1 dose of oral cladribine, followed by 4 daily doses of cladribine by vein
  Interventions: Drug: Cladribine
- Cohort 2 (PK) (Experimental): Participants will only receive 1 dose of oral cladribine, followed by 4 daily doses of cladribine by vein
  Interventions: Drug: Cladribine
- Cohort 3 (All-Oral HCL) (Experimental): Participants will all receive the same dose of oral cladribine over the course of 5 days.
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — Given by PO and Given by IV (vein)
  Other Names: Leustatin®; 2-CdA

SUMMARY:
To compare an investigational oral form of the drug cladribine to the FDA approved form of the drug when it is given by vein (IV).

DETAILED DESCRIPTION:
Objectives:

* To compare the pharmacokinetic (PK) properties of oral cladribine (investigational product) and intravenous (IV) cladribine (reference standard drug) when administered to patients with hairy-cell leukemia (HCL) or T-cell prolymphocytic leukemia (T-PLL).

Primary:

* To identify a dose of oral cladribine that is bioequivalent to IV cladribine when the IV dose is administered via a 2-hour infusion to patients with HCL or T-PLL. Area under the curve (AUC) and maximum concentration (Cmax) will be measured and relative exposure of oral and IV cladribine will be assessed based on the geometric mean ratio and associated 90% confidence interval for dose-normalized AUCs and Cmax for oral-to-IV cladribine, as estimated from an appropriate linear mixed effects model.

Secondary:

* To assess the plasma PK of oral cladribine following single-dose and multiple-dose administration.
* To identify a dose of oral cladribine that provides comparable exposure (AUC) to IV cladribine when the IV dose is administered via a 2-hour infusion to patients with HCL or T-PLL.
* To assess the safety of oral cladribine in patients with HCL or T PLL. No formal efficacy evaluations will be performed in this study. All patients will be observed for complete remission (CR), complete remission without minimal residual disease (MRD), partial response (PR), progressive disease (PD) or stable disease (SD) at the end of the study, although response is not a study endpoint.

ELIGIBILITY:
Inclusion Criteria:

Study participants must meet the following inclusion criteria

1. Patients, both men and women of all races and ethnic groups, aged ≥ 18 years are eligible for enrollment.
2. Provision of written informed consent prior to any study related procedures.
3. Patients with newly diagnosed or previously treated HCL who have indication for therapy and are candidates for cladribine therapy (all 3 cohorts).
4. Patients with previously treated T-cell prolymphocytic leukemia who have received at least one course of alemtuzumab-based treatment, who have documented indication for therapy and who are candidates for cladribine therapy (Cohort 1 and 2) only.
5. Adequate renal and hepatic organ function as indicated by the following laboratory values:

   1. Creatinine clearance ≥ 60 mL/min
   2. Serum total bilirubin ≤1.5×ULN (with the exception of patients with known Gilbert's syndrome: serum total bilirubin must be <3×ULN in these patients)
   3. Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and alanine aminotransferase (serum glutamic pyruvic transaminase) ≤2.5×ULN or ≤5×ULN if due to leukemic involvement).
6. Adequate cardiac function with a left ventricular ejection fraction ≥45%.
7. Female patients are eligible to enter and participate in the study if they are of non-childbearing potential. Female patients of childbearing age must have a negative pregnancy test at screening and must not be breastfeeding and also agree to use at least 2 forms of effective birth control during the study treatment period and for at least 3 months after the last dose of investigational product. (See definitions in Appendix 2)
8. Male patients are eligible to enter and participate in the study if they agree to use effective methods of contraception during the study treatment period and for at least 3 months after the last dose of investigational product. (See definitions in Appendix 2)

Exclusion Criteria:

Study participants must not meet any of the following study exclusion criteria:

1. Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, malabsorption, or psychiatric illness/social situations that would limit compliance with study requirements.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the compounds in the study.
3. Receipt of live or live-attenuated vaccines within 4-6 weeks preceding oral cladribine treatment, planned during cladribine treatment or after cladribine treatment until the participant's immune system is no longer weakened (e.g., white blood cell counts are within normal limits).
4. Active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody at screening. Patients who are hepatitis C antibody positive will need to have a negative PCR result prior to enrollment. Those who are hepatitis C PCR positive will be excluded. Patients who are hepatitis B virus surface antigen positive or hepatitis B PCR positive will be excluded. Patients who are anti-HBc antibody positive and who are surface antigen negative will need to have a negative PCR result before enrollment.
5. Human immunodeficiency virus (HIV) positive with a viral load >400 copies/mL and a CD4+ T-cell count of <350 cells/µL or with a history of an acquired immunodeficiency syndrome (AIDS) opportunistic infection within the past 12 months.
6. Legal incapacity or limited legal capacity.
7. Inability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation.
8. Patients unwilling to comply with protocol requirements related to the assigned cohort.
9. Patients with baseline QTc >470 msec will not be enrolled in Cohort 1. If QTc changes are observed in response to cladribine in Cohort 1, then the protocol will be amended to exclude patients with baseline QTc >470 msec from Cohorts 2 and 3, as well

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org